CLINICAL TRIAL: NCT05125822
Title: Adaptive Mechanisms Responsible for Weight Change in Youth With Obesity
Acronym: ADMIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PEDS-2021-30024; STUDY00014425 (Other: University of Minnesota HRPP)
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: This is a single group study that will consist of two interventions: an 8-week meal replacement therapy period in which participants are asked to reduce their body mass index (BMI) by >/= 5% by following a prescribed eating regimen and standardized lifestyle/behavior modification counseling which will occur every 2 weeks throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meal Replacement and Lifestyle Therapy (Experimental): Participants in this study will have an 8-week meal replacement therapy period in which they are asked to reduce their BMI by 5% by following a prescribed eating regimen consisting of meal replacement shakes and/or frozen meals for breakfast and lunch. For dinner they will consume a pre-packaged frozen entree to be consumed with two servings of fruit and three servings of vegetables per day. Participants will also have lifestyle/behavioral modification counseling every 2 weeks throughout the entire study.
  Interventions: Other: Meal replacement and lifestyle modification

INTERVENTIONS:
Other: Meal replacement and lifestyle modification — Meal replacement and lifestyle modification

SUMMARY:
In this study, doctors want to find out more about why people who lose weight often regain the weight that they have lost once they resume a regular diet and whether hormones might play a role in weight regain. The study is divided into two parts, called the meal replacement period and the follow-up period. The meal replacement period will consist of drinking a shake for breakfast and lunch and eating a frozen meal for dinner that is calorie controlled. Individuals will also be asked to eat two servings of fruit and three servings of vegetables each day. The study will provide the shakes and the frozen entrees, participants are asked to supply the fruits and vegetables.

Participation in this study will last for up to 35 weeks. There will be 10 in-person visits and 13 visits by phone or over Zoom over the 35 weeks.

DETAILED DESCRIPTION:
Individuals who are found to be eligible to participate will have two study interventions: An 8-week meal replacement therapy period in which they are asked to reduce their BMI by >5%. Participants will be asked to strictly follow the individually-prescribed eating regimen which will include meal replacement shakes and/or frozen meals to be used for breakfast and lunch. For dinner, the study will provide pre-packaged frozen entrée meals to be consumed with two servings of fruit and three servings of vegetables per day. Meal replacement compliance will be assessed by requiring participants to maintain a dietary log throughout the study. The percentage of days for which the protocol was followed (no additional calories consumed) will serve as the primary metric of compliance.

Participants will also receive a standardized lifestyle/behavioral modification counseling every 2 weeks throughout the entire study, which will be delivered at each in-person study visit and via virtual platform of phone when there is no in-person study visit scheduled. The lifestyle curriculum will incorporate evidence-based behavior change principles including dietary modification, energy expenditure modification, behavior modification and family involvement and support. To ensure fidelity and adherence to the delivery protocol, a manual will be developed for each session that trained staff will follow when administering the curriculum.

ELIGIBILITY:
Inclusion Criteria:

* 11 to less than 16 years old
* BMI > 30 kg/m^2 or 95th BMI percentile
* Tanner stage 2, 3, or 4

Exclusion Criteria:

* Tanner stage 1 and 5
* Prior bariatric surgery
* Current or recent (< 3 months prior to enrollment) use of anti-obesity medication(s) defined as orlistat, metformin, phentermine, topiramate, combination phentermine/topiramate, liraglutide, and/or combination naltrexone/bupropion (monotherapy use of naltrexone or bupropion is not an exclusion)
* Monogenic and hypothalamic obesity
* Polycystic ovary syndrome (diagnosed by a physician)
* Pregnancy or planned pregnancy
* Current use of supplemental hormones
* Individuals with a diagnosed eating disorder of anorexia nervosa, bulimia or binge eating disorder
* Type 1 or 2 diabetes
* Treatment with growth hormones
* Thyroid disease/problem
* Has had cancer in the last 10 years

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Estimated)
Dates: Start 2023-08-26 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in fat mass regain after initial weight loss with meal replacement therapy (MRT) | 17 weeks.
  We hypothesize that the greater the initial weight loss with MRT the greater the fat mass regain at 26 weeks.
Change in ghrelin | 17 weeks.
  We hypothesize that after the initial weight loss with MRT that we will see an increase in the level of the appetite regulating hormone ghrelin.
Change in gastric inhibitory polypeptide | 17 weeks
  We hypothesize that after the initial weight loss with MRT that we will see an increase in the level of the appetite regulating hormone gastric inhibitory polypeptide.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Ryder, PhD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided